CLINICAL TRIAL: NCT05246631
Title: Haloperidol Compared to Dexamethasone in Lowering Postoperative Nausea and Vomiting and Pain in Adult After Laparoscopy
Brief Title: Haloperidol and Dexamethasone Towards Postoperative Nausea and Pain in Adult After Laparoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Aldy Heriwardito, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IndonesiaUAnes393
Record Dates: First submitted 2022-01-25; First posted 2022-02-18 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Laparoscopy; Postoperative Nausea and Vomiting
Keywords: dexamethasone; haloperidol; nausea; pain; vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Nausea; Pain; Vomiting | interventions — Calcium Dobesilate; Dexamethasone; Haloperidol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dexamethasone (Active Comparator): 5 mg intravenous dexamethasone
  Interventions: Drug: Dexamethasone injection
- Haloperidol (Active Comparator): 1 mg intravenous haloperidol
  Interventions: Drug: Haloperidol Injection

INTERVENTIONS:
Drug: Dexamethasone injection — Group A consisted of patients given 5 mg intravenous dexamethasone after induction.
  Other Names: dexamethasone
  Arms: Dexamethasone
Drug: Haloperidol Injection — Group B consisted of patients given 1 mg intravenous haloperidol one hour before the surgery ended
  Other Names: haloperidol
  Arms: Haloperidol

SUMMARY:
This study aim to find out the effectiveness of 1 mg intravenous haloperidol compared to 5 mg intravenous dexamethasone to prevent the occurrence of nausea and vomiting also as pain control in adult patients after laparoscopic surgery.

DETAILED DESCRIPTION:
Eighty subjects (n=40 for each group) scheduled for laparoscopic-assisted surgery were enrolled in a randomized double-blind clinical trial. One milligram intravenous haloperidol was given one hour before the end of surgery, while 5 mg intravenous dexamethasone was given right after induction. The occurrence of Postoperative Nausea and Vomiting (PONV) and visual analog scale (VAS) pain score were recorded.

ELIGIBILITY:
Inclusion Criteria:

* underwent laparoscopic surgery (gynecology, digestive, or urology surgery)
* American Society of Anesthesiologist (ASA) physical status 1-3

Exclusion Criteria:

* psychological or neurological disorders (routine haloperidol consumption)
* history of allergic reaction to dexamethasone or haloperidol
* diabetes mellitus
* did not give the consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Nausea and Vomiting | Within 24 hours postoperative
  Number of patients experiencing nausea and vomiting postoperative

SECONDARY OUTCOMES:
Pain and VAS | 0-2 hours, 2-6 hours, 6-12 hours, and 12-24 hours postoperative
  Visual Analog Scale (VAS) score, the minimum score is 0 and the maximum score is 10. The higher scores mean a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Aldy Heriwardito, Doctor, Principal Investigator — Indonesia University
Locations (1):
- Cipto Mangunkusumo Central National Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided